CLINICAL TRIAL: NCT04184167
Title: Role of Intermittent Fasting Before Intracytoplasmic Sperm Injection
Brief Title: Role of Intermittent Fasting Before ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Role of intermittent fasting
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent fasting (Active Comparator): intermittent fasting before ICSI
  Interventions: Other: intermittent fasting 4 months before ICSI
- No intermittent fasting (Placebo Comparator): Usual diet
  Interventions: Other: intermittent fasting 4 months before ICSI

INTERVENTIONS:
Other: intermittent fasting 4 months before ICSI — women will start intermittent fasting before starting ICSI by 4 months

SUMMARY:
intermittent fasting could have a role in infertility

DETAILED DESCRIPTION:
intermittent fasting could have a role in infertility and could adjust the body weight before ICSI

ELIGIBILITY:
Inclusion Criteria:

* women with infertility

Exclusion Criteria:

* ovarian factor or uterine factor of infertility

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertile women
Enrollment: 100 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-09-02 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
the number of women who will have positive pregnancy test after ICSI | within 6 months
  The women who will get pregnant after ICSI with positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (2):
- Egypt (2):
  - Algazeerah and helwan university, Giza
  - Algazeerah, Giza